CLINICAL TRIAL: NCT05997927
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of VC005 Tablets in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Clinical Study of VC005 Tablets in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-202
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VC005 Tablets Low Dose groups (Experimental)
  Interventions: Drug: VC005 tablets; Drug: VC005 Tablets Placebo
- VC005 Tablets Medium Dose groups (Experimental)
  Interventions: Drug: VC005 tablets; Drug: VC005 Tablets Placebo
- VC005 Tablets High Dose groups (Experimental)
  Interventions: Drug: VC005 tablets; Drug: VC005 Tablets Placebo
- VC005 Tablets Placebo groups (Placebo Comparator)
  Interventions: Drug: VC005 Tablets Placebo

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 12 weeks
  Arms: VC005 Tablets High Dose groups; VC005 Tablets Low Dose groups; VC005 Tablets Medium Dose groups
Drug: VC005 Tablets Placebo — VC005 placebo groups repeat administration for 12 weeks

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, controlled phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient understands and voluntarily signs the Informed Consent Form (ICF), and has the willingness and ability to complete the regular visits, treatment plans, laboratory tests and other experimental procedures required by the program.
2. Male or female patients aged ≥18 and ≤75 years at the time of signing the ICF.
3. Meet Hanifin-Rajka diagnostic criteria at screening and have atopic dermatitis （AD) symptoms for at least 1 year prior to baseline.
4. At screening and baseline, meets criteria for moderately severe AD based on the investigator's assessment of 3 of the following:Eczema area and severity index (EASI) score ≥12;Psoriasis Area Severity Index (IGA) score ≥3;AD involvement in ≥10% of the Body Surface Area (BSA).
5. Recent (within 1 year prior to screening) topical treatment for AD with inadequate or intolerant clinical response, as determined by the investigator.
6. Able and willing to use only stabilized doses of emollients that do not contain ingredients that interfere with the evaluation of efficacy, uniformly provided by the Sponsor, beginning at least 7 days prior to Baseline and continuing for the duration of the study.
7. Non-lactating female patients of child-bearing potential (WOCBP) who have a negative pregnancy test at Screening and who are committed to adequate and effective contraception or abstinence for the duration of the study as well as for 28 days after completion of treatment with the investigational medicinal product.
8. Male patients commit to use adequate and effective contraception or abstinence for the duration of the study and for 28 days after completion of treatment with the investigational drug. In addition, male patients must agree that they will not donate sperm during this period.

Exclusion Criteria:

-

1. Presence of the following diseases or history of disease:

1. Inability to swallow the test drug or refractory nausea and vomiting, malabsorption, extracorporeal biliary shunt, or the presence of a gastrointestinal disorder (e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome) or other malabsorption condition that interferes with the absorption of the drug;
2. Current or history of lymphoproliferative disorders or presence of signs or symptoms suggestive of possible lymphoproliferative disorders of lymphoid tissue, including lymphadenopathy or splenomegaly; malignancies of any kind, or a history of any malignancy within the 5 years prior to Screening (except for completely resected carcinoma in situ of the cervix or non-metastatic squamous cell or basal cell carcinoma of the skin or papillary carcinoma of the thyroid gland);
3. Patients with prior thromboembolism (including deep vein thrombosis, pulmonary embolism, arterial thrombosis, etc.) or other high-risk groups prone to thromboembolism;
4. Patients with a history of herpes virus infection within the last 1 month or those with recurrent episodes of herpes zoster (≥2), disseminated herpes zoster, disseminated herpes simplex, or those for whom herpes zoster or herpes simplex infections cannot be excluded at this time;
5. History of any persistent or chronic infection at screening or prior to randomization (e.g., chronic pyelonephritis, chronic bronchitis) or presence of other infections judged unsuitable for enrollment in this study by the investigator; history of deep interstitial/tissue infections (e.g., fasciitis, abscess, osteomyelitis) within 12 months prior to baseline; history of conditionally causative bacterial infections (e.g., cytomegalovirus infections, pulmonary Aspergillosis, etc.); history of hospitalized infections (viral, bacterial, fungal, parasitic, etc.) within 3 months prior to baseline;
6. Immunodeficiency diseases or first-degree relatives with hereditary immunodeficiency diseases; etc.

2. Any one of the laboratory test indicators at the screening test meets the following criteria:

(1) White blood cell count (WBC) <3×109/L, absolute neutrophil count (ANC) <1.5×109/L, absolute lymphocyte count (ALC) <0.8×109/L, platelet (PLT) <100×109/L, hemoglobin (Hb) <90 g/L; etc; 3. Being on/taking or have a history of the following treatments/medications:

1. Use of systemic anti-infective drugs within 14 days prior to baseline;
2. Use of any AD topical therapy, including but not limited to topical corticosteroid (TCS), topical calcineurin inhibitors (TCI), phosphodiesterase (PDE) inhibitors,Janus kinase inhibitors, within 2 weeks prior to baseline;
3. Use of any kind of systemic systemic therapy for AD, including but not limited to immunosuppressants, corticosteroids, phosphodiesterase 4 (PDE4) inhibitors, and participation in other interventional clinical trials with an indication of AD within 4 weeks (or 5 t1/2, whichever is longer) prior to Baseline;
4. Subjects with a positive test result on the gamma-interferon (IFN-γ) release assay (QUANTIFERON®-TB GOLD or T-SPOT.TB®) at Screening, with the exception of those who, in the judgment of the Investigator, require prophylaxis and have been on prophylaxis for ≥ 4 weeks.

5. Substantial blood loss, receipt of blood transfusion, or blood donation (≥400 mL) within 3 months prior to baseline.

6、 Known or suspected allergy to the main components and excipients of VC005 or similar drugs.

7. Women who are planning to become pregnant, pregnant or breastfeeding. 8, History of alcohol abuse [>14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine)] in the 6 months prior to baseline that cannot be stopped during the trial.

9. Patients who, in the judgment of the investigator, have other reasons that make them unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in EASI score | week 12
  Percentage change from baseline in EASI score at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Chinese Academy of Medical Sciences Hospital of Skin Disease
Locations (1):
- Chinese Academy of Medical Sciences Hospital for Skin Diseases, Nanjing, Jiangsu, China